CLINICAL TRIAL: NCT06100900
Title: An Open-Label, Multicenter, Intra-Subject Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Therapeutic Potential of BCX10013 in Subjects with Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Dose Escalation of BCX10013 in Participants with Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCX10013-105
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria; Factor D; complement inhibitor; alternative pathway inhibitor; BioCryst
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Intervention Model Description: Multiple dose levels of BCX10013 are planned for escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCX10013 (Experimental): Participants with PNH will receive BCX10013 daily for 4 weeks before dose escalation may occur.
  Interventions: Drug: BCX10013

INTERVENTIONS:
Drug: BCX10013 — Multiple dose levels may be tested in this study.

SUMMARY:
This is a multicenter, open-label, intra-subject, dose escalation study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and therapeutic potential of BCX10013 in participants with PNH. Approximately 8 participants will be enrolled in this study. Participants may receive treatment for up to 52 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or non-pregnant, non-lactating female adults ≥ 18 years old.
2. Documented diagnosis of PNH confirmed by flow cytometry.
3. Body mass index (BMI) ≤ 40 kg/m^2.
4. Are either: (a) naïve to treatment with a complement inhibitor; or (b) have received no treatment with ravulizumab for at least 12 months prior to the screening visit and have received no treatment with eculizumab or pegcetacoplan for 6 months prior to the screening visit.
5. Documentation of current vaccinations against N. meningitidis, S. pneumoniae, and H. influenzae type B [Hib] or willingness to start vaccination series at least 14 days prior to Day 1.

Key Exclusion Criteria:

1. Known history of or existing diagnosis of hereditary complement deficiency.
2. History of hematopoietic cell transplant or solid organ transplant or anticipated candidate for transplantation during the study.
3. Myocardial infarction or cerebrovascular accident within 30 days prior to screening, or current and uncontrolled clinically significant cardiovascular or cerebrovascular condition, including unstable angina, severe congestive heart failure, unexplained syncope, arrhythmia, and critical aortic stenosis.
4. History of malignancy within 5 years prior to the screening visit.
5. Treatment with anti-thymocyte globulin within 180 days prior to the screening visit.
6. Initiation of treatment with an erythropoiesis-stimulating agent (eg, erythropoietin), a thrombopoietin receptor agonist (eg, eltrombopag), or danazol within 28 days prior to the screening visit.
7. Receiving iron with an unstable dose (ie, increasing or decreasing) in the 28 days prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Graded Laboratory Abnormalities, and Changes From Baseline (CFB) in Laboratory Analytes, Vital signs, Electrocardiograms (ECGs), and Physical Examination Findings. | up to 52 weeks

SECONDARY OUTCOMES:
CFB in Lactate Dehydrogenase | Baseline, Week 52
CFB in the Ratio of Total PNH Red Blood Cell Clone Size to PNH White Blood Cell Clone Size | Baseline, Week 52
CFB in Hemoglobin | Baseline, Week 52
Percentage of Participants who are Transfusion-free | 52 weeks
Percentage of Participants Achieving a Within-subject Clinically Meaningful CFB in the FACIT-Fatigue scale | 52 weeks
CFB in Other Clinical Biomarkers of PNH Disease Activity including absolute reticulocyte count, total PNH red blood cell clone size, haptoglobin levels, total bilirubin, and aspartate transaminase | Baseline, Week 52
Number of Participants with Clinical PNH Symptoms | up to 52 weeks
Concentration of BCX10013 and its Metabolite(s) in Plasma | Pre-dose, 0.5, 1, 2, 4, and 6 hours post dose on Day 1, Week 2, and Week 4
Concentration of BCX10013 and its Metabolite(s) in Urine (if applicable) | Pre-dose and all urine from 0 to 6 hours post dose on Day 1, Week 2, and Week 4

CONTACTS AND LOCATIONS:
Locations (4):
- BioCryst Investigative Site, Ampang, Malaysia
- South Africa (3):
  - BioCryst Investigative Site, Bloemfontein
  - BioCryst Investigative Site, Cape Town
  - BioCryst Investigative Site, Pretoria

IPD SHARING:
Plan to Share IPD: No